CLINICAL TRIAL: NCT03484013
Title: Totally Percutaneous Approach to Endovascular Treatment of Aortic Aneurysms (PEVAR-PRO)
Acronym: PEVAR-PRO
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: PEVAR-PRO/141/OSR
Record Dates: First submitted 2017-12-12; First posted 2018-03-30 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Aneurysm; Aneurysm Abdominal; Aneurysm Thoracic; Aneurysm, Thoracoabdominal Aortic
MeSH Terms: conditions — Aneurysm; Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic; Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Purpose of the study is the evaluation of the applicability of the percutaneous technique through double Proglide and Pre-Close Technique to the treatment of complex aortic aneurysms with thoracic endoprosthesis (TEVAR), fenestrated or branched (F / B-EVAR) in which patient-related factors, the devices used or the procedure, could affect the performance.

DETAILED DESCRIPTION:
Endovascular treatment using a percutaneous technique (Percutaneous Endovascular Aneurism Repair - P-EVAR) has been used with increasing frequency to treat aortic aneurysms by reducing operative times, postoperative pain and length of stay, compared to treatment by surgical femoral access. During EVAR procedures, two accesses to the femoral arteries are required to introduce the necessary tools for the stentgraft implantation. Such accesses can be classically obtained by surgical incision, isolation of the common femoral arteries and direct introduction of the devices.

Alternatively, the most modern approach involves direct puncture of the artery (without the need for incision), through the skin and closure of the arterial breach through prolonged manual compression of the vascular closure or systems (Vascular Closure Devices - VCD) specifically designed. Among the various closure devices one of the most used and studied is the Perclose Proglide (Abbott Vascular, Santa Clara CA, USA) that allows to affix a polypropylene stitch to close the arterial breach. When closing high-caliber accesses (> 8 French) it is necessary to use two devices that must be positioned before inserting the introducer ("Pre-Close Technique").

Few studies have so far evaluated the application of this method to the treatment of complex cases such as thoracic or thoracoabdominal aortic aneurysms that requiring the use of high caliber introducers.

The objective of the study is the evaluation of the technical success and clinical outcomes of the PEVAR technique with a double vascular suture device Perclose ProGlide (Abbott Illinois, U.S.A.).Endovascular treatment using a percutaneous technique (Percutaneous Endovascular Aneurism Repair - P-EVAR) has been used with increasing frequency to treat aortic aneurysms by reducing operative times, postoperative pain and length of stay, compared to treatment by surgical femoral access. During EVAR procedures, two accesses to the femoral arteries are required to introduce the necessary tools for the stentgraft implantation. Such accesses can be classically obtained by surgical incision, isolation of the common femoral arteries and direct introduction of the devices.

Alternatively, the most modern approach involves direct puncture of the artery (without the need for incision), through the skin and closure of the arterial breach through prolonged manual compression of the vascular closure or systems (Vascular Closure Devices - VCD) specifically designed. Among the various closure devices one of the most used and studied is the Perclose Proglide (Abbott Vascular, Santa Clara CA, USA) that allows to affix a polypropylene stitch to close the arterial breach. When closing high-caliber accesses (> 8 French) it is necessary to use two devices that must be positioned before inserting the introducer ("Pre-Close Technique").

Few studies have so far evaluated the application of this method to the treatment of complex cases such as thoracic or thoracoabdominal aortic aneurysms that requiring the use of high caliber introducers.

The objective of the study is the evaluation of the technical success and clinical outcomes of the PEVAR technique with a double vascular suture device Perclose ProGlide (Abbott Illinois, U.S.A.).

This is a retrospective observational study (320 cases treated in San Raffaele hospital in Milan, during the period: October 2015 - 31 December 2019).

The chronology of the assessments will include:

* An immediate evaluation at the end of the procedure by performing the ecocolordoppler examination of the percutaneous accesses performed (as per routine). On the basis of longitudinal and sagittal scans of the vessel, the Physician must check the presence of the above complications that could be considered as "failure" of percutaneous access. In the event that these complications are clinically evident (eg uncontrollable bleeding from the puncture site), in the interest of a prompt management of the surgical problem, it will not be necessary to perform an ecocolordoppler examination and the outcome will be assigned "failure ".
* A second echocolordoppler assessment performed on the first postoperative day (as per routine) The study will be conducted in accordance with the ethical principles deriving from the Helsinki Declaration and the current legislation on Observational Studies.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged ≥ 18 years, belonging to the Operative Unit of Vascular Surgery of the San Raffaele Hospital,
* patients candidates for endovascular treatment for thoracic, thoracoabdominal or abdominal aortic pathologies.

Exclusion Criteria:

- There are no criteria for exclusion of subjects from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: a sample of 320 subjects will be analyzed (considering the cases treated in the period: October 2015 - 31 december 2019).
  The analysis of the retrospective data, will be based on the consultation of the archive of the individual treated patients, present on software platform belonging to the San Raffaele Hospital Information System) as well as the medical records.
  An informatic database will be set up for the exclusive use of investigators. The data will be analyzed subsequently through the application of descriptive and inferential statistics techniques.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
technical success | during the surgery
  Use of femoral artery access in endovascular repair of aortic aneurysm (time frame between 2015 and 2020)
  * Endovascular procedure: TEVAR - EVAR - B/FEVAR
  * Side of femoral access: right- left
  * Employment of downsizing on the femoral access: yes - no, as reported on patients' charts and operative report
  * Size of percutaneous access sheath employed measured in French - Fr
  * Number of percutaneous access vessel closure devices employed
  * Access closure specific outcome: success - failure, as reported on patients' charts and operative report
  * Cause of failure: hemorrhagic - occlusive, as reported on patients' charts and operative report

SECONDARY OUTCOMES:
minor complications | 30 days after surgery
  Femoral access vascular anatomy and patient's characteristics (time frame between 2015 and 2020):
  * Previous surgical access to ipsilateral femoral artery: yes - no
  * Previous deployment of percutaneous vascular closure devices to ipsilateral femoral artery: yes - no
  * Diameter of femoral artery measured in millimiters (mm)
  * Presence of calcification at access site: less or equal to1/3 of circumference - between 1/3 (excluded) and 2/3 (included) - more than 2/3 as measured on preoperative CT scan
  * Localization of calcification: anterior - posterior - circumferential - lateral
  * Body mass index reported as bare number defined as weight (kg)/height^2(m^2)

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

REFERENCES:
- [Derived] Melloni A, Grandi A, Spelta S, Salvati S, Loschi D, Lembo R, Melissano G, Chiesa R, Bertoglio L. Outcomes of routine use of percutaneous access with large-bore introducer sheaths (>21F outer diameter) during endovascular aneurysm repair. J Vasc Surg. 2021 Jan;73(1):81-91. doi: 10.1016/j.jvs.2020.04.504. Epub 2020 May 19. PMID 32442603